CLINICAL TRIAL: NCT04610333
Title: On Top of Everything. A Study Protocol for a Cluster-Randomised Controlled Trial Testing a Teacher Training Programme to Teach Mindfulness Among Students in Danish Upper Secondary Schools and Schools of Health and Social Care
Brief Title: On Top of Everything
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15092020
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2020-09

CONDITIONS: Mental Health; Youth; Mindfulness; Stress
Keywords: School-based intervention; Population-based preventive strategy; Public health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School teacher training (Experimental): Teacher training programme:
  * MBSR according to international standards (2.5 hours group session once a week in 8 weeks; a silence retreat day; and 45-60 minutes homework six days a week). Content in accordance with MBSR curriculum.
  * Four-day residental course
  * 3 x 2 seminar days
  Modified MBSR programme delivered to the students:
  - 1hour group session once a week in 10 weeks taught by the educated teachers on class
  Interventions: Behavioral: Modified MBSR programme
- Usual practice (No Intervention)

INTERVENTIONS:
Behavioral: Modified MBSR programme — 1 hour group session once a week in 10 weeks
  Arms: School teacher training

SUMMARY:
Our primary aim of this trial is to evaluate the effectiveness of a teacher training programme to teach mindfulness as part of regular classroom teaching in the total population of students in Danish upper secondary schools and schools of health and social care, respectively, on students' self-reported mental health at six-month follow-up.

Our secondary aim is to evaluate the effectiveness of the teacher training programme to teach mindfulness in a vulnerable subgroup of students on their self-reported mental health at three and six months after baseline.

DETAILED DESCRIPTION:
The study is designed as a pragmatic cluster randomised two-arm trial including 43 Danish schools (30 upper secondary schools and 13 schools of health and social care). The schools included a total of 76 school teachers for teacher training (44 teachers from upper secondary schools and 32 teachers from schools of health and social care). Each included teacher will be asked to recruit a class of students (15-30 students) to test the effectiveness of the modified MBSR programme (in total approx. 1.000 students).

ELIGIBILITY:
Inclusion Criteria:

* All students in the enrolled school classes

Exclusion Criteria:

* None

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 992 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Warwick-Edinburgh Mental Well-Being Scale (SWEMWBS) - The short version | Six months after baseline
  Change in the score among the total study population

SECONDARY OUTCOMES:
Warwick-Edinburgh Mental Well-Being Scale (SWEMWBS) - The short version | Three months after baseline
  Change in the score among the total study population
Strengths and Difficulties Questionnaire (SDQ) - The youth self-report version | Three months after baseline
  Change in the score among the total study population
Strengths and Difficulties Questionnaire (SDQ) - The youth self-report version | Six months after baseline
  Change in the score among the total study population
Perseived Stress Scale | Three months after baseline
  Change in the score among the total study population
Perseived Stress Scale | Six months after baseline
  Change in the score among the total study population
Depression Anxiety Stress Scale (DASS) - The short form version | Three months after baseline
  Change in the score among the total study population
Depression Anxiety Stress Scale (DASS) - The short form version | Six months after baseline
  Change in the score among the total study population
Brief Resilience Scale (BRS) | Three months after baseline
  Change in the score among the total study population
Brief Resilience Scale (BRS) | Six months after baseline
  Change in the score among the total study population
Three-Item Loneliness Scale (T-ILS) | Three months after baseline
  Change in the score among the total study population
Three-Item Loneliness Scale (T-ILS) | Six months after baseline
  Change in the score among the total study population
Experiences Questionnaire (EQ) - Decentering subscale | Three months after baseline
  Change in the score among the total study population
Experiences Questionnaire (EQ) - Decentering subscale | Six months after baseline
  Change in the score among the total study population
EQ-5D | Three months after baseline
  Change in the score among the total study population
EQ-5D | Six months after baseline
  Change in the score among the total study population
Karolinska Sleep Questionnaire - Modified version | Three months after baseline
  Change in the score among the total study population
Karolinska Sleep Questionnaire - Modified version | Six months after baseline
  Change in the score among the total study population

CONTACTS AND LOCATIONS:
Overall Officials: Lise Juul, PhD, Principal Investigator — Danish Center for Mindfulness
Locations (1):
- Danish Center for Mindfulness, Aarhus, Brabrand, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data will be shared by reasonable request, following publication of planned papers.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Juul L, Frydenberg M, Bonde EH, Beck MS, Goetzsche K, Bruggisser S, Fjorback LO. Introducing a mindfulness-based intervention in school curriculum to 16-24-year-olds. A nationwide cluster-randomized trial. Npj Ment Health Res. 2025 Aug 11;4(1):37. doi: 10.1038/s44184-025-00150-w. PMID 40789917
- [Derived] Beck MS, Juul L, Frydenberg M, Fjorback LO. On Top of Everything: a study protocol for a cluster-randomised controlled trial testing a teacher training programme to teach mindfulness among students in Danish upper secondary schools and schools of health and social care. Trials. 2023 Jan 6;24(1):17. doi: 10.1186/s13063-022-06920-7. PMID 36609335